CLINICAL TRIAL: NCT00050466
Title: A Pilot Study Using the Dynamic Light Scattering Device (DLS) Combined With Keratoscopy on the Cornea in Vivo
Brief Title: Dynamic Light Scattering and Keratoscopy for Corneal Examination
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030012; 03-EI-0012
Record Dates: First submitted 2002-12-09; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-09

CONDITIONS: Corneal Diseases
Keywords: Normal Volunteers; Dynamic Light Scattering (DLS); Corneal Opacities; Cornea; Transparency; Vision
MeSH Terms: conditions — Corneal Diseases; Corneal Opacity

SUMMARY:
This pilot study will examine the usefulness of a new instrument called the Dynamic Light Scattering (DLS) device for documenting and monitoring changes in the cornea, the front part of the eye where contact lenses are placed. The DLS device uses a low-intensity laser similar to that used in supermarket checkouts to measure the cloudiness of the cornea. The results of this study may lead to further investigations using DLS to discover the cause of corneal clouding and to develop treatments to prevent it.

Healthy volunteers and patients with corneal clouding or opacification 18 years of age and older may be eligible for this study.

Participants will have a standard eye examination, including a check of visual acuity and eye pressure. The retina will also be examined and photographs of the cornea may be taken. For the DLS test, the subject sits in front of the device and looks at a yellow-green target while the cloudiness of the cornea is measured. Subjects will be tested four times. The entire procedure takes less than 30 minutes.

DETAILED DESCRIPTION:
Corneal disease and injuries are the leading cause of visits to eye care clinics in the US today. These diseases are also some of the most painful eye disorders. Two important areas for research on the cornea are 1) to explore and understand the molecular basis of corneal transparency and 2) to analyze the molecular nature of corneal inflammation and wound healing. We have developed a new clinical device to understand molecular changes that occur in the lens, called Dynamic Light Scattering (DLS) device. Studies have shown its potential in the detection of the earliest changes occurring in the cataract, and have also shown good test retest reproducibility of the system. We now would like to apply this technique to study changes that occur in corneal opacification. In this pilot project, we would like to study the normal cornea in young and older persons (volunteers) as well as cloudy, opaque corneas. This will allow us to determine if useful data can be obtained, and if so, lead to further studies in various corneal disorders caused by trauma, infections, and dystrophies, as well as those caused by systemic or inherited disorders.

ELIGIBILITY:
INCLUSION CRITERIA:

Individuals greater than or equal to 18 years of age.

Controls:

Control subjects must have normal, clear corneas as determined by slit lamp biomicroscopy and central corneal thickness less than 0.55 mm centrally.

Patients:

Patients with corneal clouding and opacification.

EXCLUSION CRITERIA:

To be eligible, participants must not satisfy the criterion below:

Individuals who cannot cooperate or keep still for the DLS measurements.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24
Dates: Start 2002-12; Study Completion 2005-09

CONTACTS AND LOCATIONS:
Locations (1):
- National Eye Institute (NEI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Datiles MB 3rd, Ansari RR, Reed GF. A clinical study of the human lens with a dynamic light scattering device. Exp Eye Res. 2002 Jan;74(1):93-102. doi: 10.1006/exer.2001.1106. PMID 11878822
- [Background] Benedek GB, Chylack LT Jr, Libondi T, Magnante P, Pennett M. Quantitative detection of the molecular changes associated with early cataractogenesis in the living human lens using quasielastic light scattering. Curr Eye Res. 1987 Dec;6(12):1421-32. doi: 10.3109/02713688709044506. PMID 3427992
- [Background] Thurston GM, Hayden DL, Burrows P, Clark JI, Taret VG, Kandel J, Courogen M, Peetermans JA, Bowen MS, Miller D, Sullivan KM, Storb R, Stern H, Benedek GB. Quasielastic light scattering study of the living human lens as a function of age. Curr Eye Res. 1997 Mar;16(3):197-207. doi: 10.1076/ceyr.16.3.197.15410. PMID 9088735